CLINICAL TRIAL: NCT01773928
Title: Randomized, Age-stratified, Double Blind, Controlled Phase 3 Study Comparing a Vero Cell-derived Trivalent Seasonal Influenza Vaccine Made by the Modified Manufacturing Process With Vaccine Made by the Current Manufacturing Process and a Licensed Trivalent Influenza Vaccine in Healthy Adults Aged 18 Years and Older
Brief Title: Inactivated Split Virus Seasonal Influenza Vaccine (Vero Cell-Derived)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 721104
Record Dates: First submitted 2013-01-17; First posted 2013-01-23 (Estimated); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Influenza
Keywords: Active immunization against influenza disease
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- VCIV - Modified manufacturing process (18-49 Years Old) Lot 1 (Experimental): Vero cell-derived trivalent influenza vaccine (VCIV)
  Interventions: Biological: Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- VCIV - Modified manufacturing process (18-49 Years Old) Lot 2 (Experimental): Vero cell-derived trivalent influenza vaccine (VCIV)
  Interventions: Biological: Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- VCIV - Modified manufacturing process (18-49 Years Old) Lot 3 (Experimental): Vero cell-derived trivalent influenza vaccine (VCIV)
  Interventions: Biological: Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- VCIV manufactured with current process (18-49 Years Old) (Active Comparator): Vero cell-derived trivalent influenza vaccine (VCIV)
  Interventions: Biological: VCIV manufactured with the current manufacturing process (VCIV current)
- Fluzone® (18-49 Years Old) (Active Comparator): Fluzone®, licensed trivalent influenza vaccine (TIV)
  Interventions: Biological: Fluzone®, licensed trivalent influenza vaccine (TIV)
- VCIV - Modified manufacturing process (≥50 Years Old) Lot 1 (Experimental): Vero cell-derived trivalent influenza vaccine (VCIV)
  Interventions: Biological: Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- VCIV - Modified manufacturing process (≥50 Years Old) Lot 2 (Experimental): Vero cell-derived trivalent influenza vaccine (VCIV)
  Interventions: Biological: Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- VCIV - Modified manufacturing process (≥50 Years Old) Lot 3 (Experimental): Vero cell-derived trivalent influenza vaccine (VCIV)
  Interventions: Biological: Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- Fluzone® (≥50 Years Old) (Active Comparator): Fluzone®, licensed trivalent influenza vaccine (TIV)
  Interventions: Biological: Fluzone®, licensed trivalent influenza vaccine (TIV)

INTERVENTIONS:
Biological: Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
  Arms: VCIV - Modified manufacturing process (18-49 Years Old) Lot 1; VCIV - Modified manufacturing process (18-49 Years Old) Lot 2; VCIV - Modified manufacturing process (18-49 Years Old) Lot 3; VCIV - Modified manufacturing process (≥50 Years Old) Lot 1; VCIV - Modified manufacturing process (≥50 Years Old) Lot 2; VCIV - Modified manufacturing process (≥50 Years Old) Lot 3
Biological: VCIV manufactured with the current manufacturing process (VCIV current)
  Arms: VCIV manufactured with current process (18-49 Years Old)
Biological: Fluzone®, licensed trivalent influenza vaccine (TIV)
  Arms: Fluzone® (18-49 Years Old); Fluzone® (≥50 Years Old)

SUMMARY:
The purpose of this study is to determine if a Vero cell-derived trivalent seasonal influenza vaccine produced by the modified manufacturing process:

1. induces immune responses comparable to that produced by the current manufacturing process
2. has an acceptable safety profile compared to a licensed trivalent seasonal influenza vaccine
3. demonstrates consistency of immune response among three different lots.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 to 49 years of age, inclusive, at the time of screening (for Cohort 18 to 49 years of age);
* Participant is 50 years of age, inclusive, or older at the time of screening (for Cohort 50 years of age or older);
* Participant gave written informed consent prior to study entry
* Participant is generally healthy without any significant medical risk conditions, as determined by the Investigator's clinical judgment through collection of medical history and performance of a physical examination;
* Participant is willing and able to comply with the requirements of the protocol;
* Participant agrees to keep a record of symptoms for the duration of the study;
* If female and capable of bearing children - participant has a negative urine pregnancy test at the study site, within 36 hours prior to vaccination, and agrees to employ adequate birth control measures for the duration of the study. For the purposes of this study adequate birth control measures incorporate one of the following FDA approved birth control measures for the duration of the study:

  * Hormonal types of birth control (such as implants, birth control pills, patches or other methods) or an intrauterine device, OR
  * A barrier type of birth control measure (i.e., condoms, diaphragms, cervical caps, etc.).

Exclusion Criteria:

* Participant has been vaccinated with seasonal trivalent influenza vaccine in the current season;
* Participant has an oral temperature of ≥100.4°F (≥38.0°C) on the day of vaccination in this study;
* Participant has received a live vaccine within 4 weeks, or an inactivated or subunit vaccine within 2 weeks of study entry;
* Participant with a known history of infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBsAgs) or Hepatitis C Virus (HCV);
* Participant has any medically diagnosed or suspected immune deficient condition based on medical history and physical examination as determined by the Investigator;
* Participant has an immune compromising condition or disease, or is currently undergoing a form of treatment or was undergoing a form of treatment within 30 days prior to study entry that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled corticosteroids (> 800 μg/day of beclomethasone dipropionate or equivalent), radiation treatment or other immunosuppressive or cytotoxic drugs (use of inhaled and nasal steroids will be permitted);
* Participant has a known history of Guillain Barré Syndrome, demyelinating disorders (including acute demyelinating encephalomyelitis (ADEM), Multiple Sclerosis) or convulsions;
* Participant has a history of severe allergic reactions or anaphylaxis as determined by the Investigator;
* Participant has a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating as determined by the Investigator;
* Participant has received any blood products (e.g. blood transfusion or immunoglobulins) within 90 days prior to study entry;
* Participant has donated one or more units of blood (approximately 450 mL) or plasma within 30 days prior to study entry;
* Participant has a functional or surgical asplenia;
* Participant has a known or suspected problem with alcohol or drug abuse as determined by the Investigator;
* Participant is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie., children, partner/spouse, siblings, parents) as well as employees of the Investigator or study site personnel conducting the study;
* If female, participant is pregnant or lactating at the time of study enrollment;
* Participant is currently enrolled or has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to study enrolment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study;
* Participant has any condition that in the opinion of the Investigator would interfere with evaluation of the vaccine or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1928 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirjhar Chatterjee, MD, Study Director — Baxter Healthcare Corporation
Locations (20):
- United States (20):
  - East Valley Family Physicians, PLC, Chandler, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Center for Clinical Trials, LLC, Paramount, California
  - California Research Foundation, San Diego, California
  - Benchmark Research San Francisco, San Francisco, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Miami Research Associates, South Miami, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Heartland Research Associates, LLC, Wichita, Kansas
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Rochester Clinical Research Inc., Rochester, New York
  - PMG Research of Cary, LLC, Cary, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Benchmark Research Austin, Austin, Texas
  - Benchmark Research, Fort Worth, Texas
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Background] StatXact 7 PROCs for SAS Users, Cytel Inc, Cambridge, 2005.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the U.S. at 20 study sites. The first participant was enrolled in January 2013.
Pre-assignment Details: 1,928 potential participants were enrolled at clinical study sites in the United States. 75 were screen failures; and 52 were not assigned to a treatment group once the randomization goals were reached. Therefore, 1,801 participants were randomized.
Groups:
- VCIV Current Process (18-49 Years Old): Vero cell-derived trivalent influenza vaccine (VCIV)
  VCIV manufactured with the current manufacturing process (VCIV current)
- VCIV - Modified Process (18-49 Years Old) Lot 1; VCIV - Modified Process (18-49 Years Old) Lot 2; VCIV - Modified Process (18-49 Years Old) Lot 3; VCIV - Modified Process (≥50 Years Old) Lot 1; VCIV - Modified Process (≥50 Years Old) Lot 2; VCIV - Modified Process (≥50 Years Old) Lot 3: Vero cell-derived trivalent influenza vaccine (VCIV)
  Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
Period: Overall Study
Arm/Group | Fluzone® (18-49 Years Old) | VCIV Current Process (18-49 Years Old) | VCIV - Modified Process (18-49 Years Old) Lot 1 | VCIV - Modified Process (18-49 Years Old) Lot 2 | VCIV - Modified Process (18-49 Years Old) Lot 3 | Fluzone® (≥50 Years Old) | VCIV - Modified Process (≥50 Years Old) Lot 1 | VCIV - Modified Process (≥50 Years Old) Lot 2 | VCIV - Modified Process (≥50 Years Old) Lot 3
Started | 201 | 201 | 200 | 200 | 200 | 204 | 199 | 197 | 199
Completed | 196 | 196 | 196 | 194 | 192 | 202 | 199 | 196 | 197
Not Completed | 5 | 5 | 4 | 6 | 8 | 2 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 4 | 4 | 7 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Subject misrepresented age | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject met exclusion criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Randomized, had to leave, never returned | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Refused vaccine, withdrew consent | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Groups:
- VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 1; VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 2; VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 3; VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1; VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 2; VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 3: Vero cell-derived trivalent influenza vaccine (VCIV)
  Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- VCIV Manufactured With Current Process (18-49 Years Old): Vero cell-derived trivalent influenza vaccine (VCIV)
  VCIV manufactured with the current manufacturing process (VCIV current)
- Total: Total of all reporting groups
Arm/Group | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 1 | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 2 | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 3 | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1 | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 2 | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 3 | Fluzone® (≥50 Years Old) | Total
Number analyzed (Participants) | 200 | 199 | 199 | 201 | 201 | 199 | 197 | 198 | 203 | 1797
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (9.09) | 34.2 (9.26) | 32.6 (9.05) | 34.4 (9.28) | 34.0 (9.28) | 61.5 (8.44) | 62.2 (8.55) | 61.5 (7.91) | 62.4 (8.71) | 46.1 (16.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 121 | 102 | 111 | 117 | 116 | 92 | 103 | 115 | 998
  Male | 79 | 78 | 97 | 90 | 84 | 83 | 105 | 95 | 88 | 799
Region of Enrollment [Number; unit: participants]
  United States | 200 | 199 | 199 | 201 | 201 | 199 | 197 | 198 | 203 | 1797

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition Antibody (HIA) Titer for Each of the Three Antigens Contained in the Vaccine
Description: Hemagglutination Inhibition Antibody (HIA) Titer for Each of the Three Antigens Contained in the Vaccine
  Two co-primary analyses relating to this primary immunogenicity outcome measure were also performed:
  Outcome Measure 2 - Noninferiority Outcome Measure 3 - Lot Consistency
Time Frame: 21 days post vaccination
Population: Immunogenicity Analysis Set. The primary immunogenicity and safety analyses groups included the VCIV Modified lots separately. The secondary immunogenicity and safety analyses groups included all three of the VCIV Modified lots pooled.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Total VCIV - Modified Process (18 - 49 Years Old) Lots 1-3; VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1; VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 2; VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 3; Total VCIV - Modified Process (≥50 Years Old) Lots 1-3: Vero cell-derived trivalent influenza vaccine (VCIV)
  Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
Arm/Group | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 1 | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 2 | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 3 | Total VCIV - Modified Process (18 - 49 Years Old) Lots 1-3 | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1 | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 2 | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 3 | Total VCIV - Modified Process (≥50 Years Old) Lots 1-3 | Fluzone® (≥50 Years Old)
Number analyzed (Participants) | 196 | 193 | 192 | 581 | 195 | 196 | 199 | 196 | 195 | 590 | 200
Titers
  Strain A/H1N1 | 269.7 [222.6 to 326.8] | 337.3 [286.9 to 396.6] | 288.5 [238.8 to 348.6] | 297.1 [267.6 to 329.8] | 264.4 [216.0 to 323.7] | 595.6 [516.9 to 686.3] | 141.3 [113.6 to 175.7] | 118.3 [93.9 to 149.1] | 112.8 [89.8 to 141.7] | 123.7 [108.6 to 140.8] | 306.3 [255.5 to 367.1]
  Strain A/H3N2 | 153.5 [127.5 to 184.9] | 245.3 [207.1 to 290.6] | 205.5 [171.1 to 246.8] | 197.5 [178.0 to 219.3] | 172.2 [144.2 to 205.6] | 314.4 [268.7 to 367.9] | 174.4 [143.6 to 211.7] | 165.8 [134.3 to 204.6] | 168.4 [135.2 to 209.6] | 169.5 [150.4 to 191.0] | 294.8 [246.7 to 352.3]
  Strain B | 86.8 [74.5 to 101.0] | 83.5 [70.7 to 98.6] | 83.6 [70.3 to 99.5] | 84.6 [77.0 to 93.0] | 60.7 [51.2 to 72.0] | 97.3 [84.3 to 112.2] | 40.5 [33.4 to 49.0] | 35.9 [29.7 to 43.4] | 30.4 [25.3 to 36.4] | 35.4 [31.7 to 39.4] | 37.1 [31.4 to 44.0]

2. Secondary Outcome: Percentage of Participants With Seroprotective Antibody Titer for Each of the Three Antigens
Description: Percentage of participants with seroprotective antibody titer [reciprocal HIA titer ≥40] for each of the three antigens contained in the vaccine
Time Frame: 21 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- VCIV - Modified Manufacturing Process (18-49 Years Old); VCIV - Modified Manufacturing Process (≥50 Years Old): Vero cell-derived trivalent influenza vaccine (VCIV)
  Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
Arm/Group | VCIV - Modified Manufacturing Process (18-49 Years Old) | VCIV - Modified Manufacturing Process (≥50 Years Old) | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | Fluzone® (≥50 Years Old)
Number analyzed (Participants) | 581 | 590 | 195 | 196 | 200
percentage of participants
  Strain A/H1N1 | 94.7 [92.5 to 96.3] | 79.0 [75.5 to 82.2] | 90.8 [85.8 to 94.4] | 100.0 [98.1 to 100.0] | 95.5 [91.6 to 97.9]
  Strain A/H3N2 | 91.6 [89.0 to 93.7] | 86.4 [83.4 to 89.1] | 90.8 [85.8 to 94.4] | 98.5 [95.6 to 99.7] | 94.0 [89.8 to 96.9]
  Strain B | 82.8 [79.5 to 85.8] | 53.6 [49.4 to 57.6] | 72.3 [65.5 to 78.5] | 88.8 [83.5 to 92.8] | 59.5 [52.3 to 66.4]

3. Secondary Outcome: Percentage of Participants Demonstrating Seroconversion to Each of the Three Antigens Contained in the Vaccine
Description: Seroconversion is defined as a ≥ 4-fold increase in HIA titer from baseline OR a reciprocal HIA titer ≥ 40 when there is no detectable HIA titer (reciprocal HIA titer < 10) at baseline
Time Frame: 21 days post vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VCIV - Modified Manufacturing Process (18-49 Years Old) | VCIV - Modified Manufacturing Process (≥50 Years Old) | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | Fluzone® (≥50 Years Old)
Number analyzed (Participants) | 581 | 590 | 195 | 196 | 200
percentage of participants
  Strain A/H1N1 | 70.9 [67.0 to 74.6] | 52.7 [48.6 to 56.8] | 64.6 [57.5 to 71.3] | 79.1 [72.7 to 84.6] | 70.5 [63.7 to 76.7]
  Strain A/H3N2 | 57.5 [53.4 to 61.5] | 50.3 [46.2 to 54.4] | 51.3 [44.0 to 58.5] | 67.9 [60.8 to 74.3] | 63.5 [56.4 to 70.2]
  Strain B | 61.4 [57.4 to 65.4] | 40.3 [36.4 to 44.4] | 54.9 [47.6 to 62.0] | 70.9 [64.0 to 77.2] | 49.0 [41.9 to 56.1]

4. Secondary Outcome: Fold Increase of HIA Titer for Each of the Three Antigens Contained in the Vaccine as Compared to Baseline
Time Frame: 21 days post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- VCIV - Modified Process (18-49 Years Old) Lots 1-3; VCIV - Modified Process (≥50 Years Old) Lots 1-3: Vero cell-derived trivalent influenza vaccine (VCIV)
  Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
Arm/Group | VCIV - Modified Process (18-49 Years Old) Lots 1-3 | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | VCIV - Modified Process (≥50 Years Old) Lots 1-3 | Fluzone® (≥50 Years Old)
Number analyzed (Participants) | 581 | 195 | 196 | 590 | 200
Titers
  Strain A/H1N1 | 9.6 [8.5 to 10.8] | 8.5 [6.8 to 10.5] | 19.9 [15.5 to 25.4] | 5.5 [4.9 to 6.2] | 12.7 [10.0 to 16.2]
  Strain A/H3N2 | 5.6 [5.0 to 6.3] | 4.8 [4.0 to 5.8] | 9.5 [7.6 to 12.0] | 5.1 [4.6 to 5.8] | 8.5 [6.8 to 10.6]
  Strain B | 6.7 [6.0 to 7.5] | 5.6 [4.7 to 6.8] | 9.1 [7.6 to 10.8] | 3.9 [3.5 to 4.3] | 4.8 [4.0 to 5.6]

5. Secondary Outcome: Percentage of Participants With Solicited Systemic Reactions
Time Frame: within 7 days post vaccination
Population: Safety Analysis Set. The primary immunogenicity and safety analyses groups included the VCIV Modified lots separately. The secondary immunogenicity and safety analyses groups included all three of the VCIV Modified lots pooled.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total VCIV - Modified Manufacturing Process (18-49 Years Old) Lots 1-3; Total VCIV - Modified Manufacturing Process (≥50 Years Old) Lots 1-3; Total VCIV - Modified Manufacturing Process (All Participants) Lots 1-3: Vero cell-derived trivalent influenza vaccine (VCIV)
  Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- Fluzone® (All Participants): Fluzone®, licensed trivalent influenza vaccine (TIV)
Arm/Group | Total VCIV - Modified Manufacturing Process (18-49 Years Old) Lots 1-3 | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | Total VCIV - Modified Manufacturing Process (≥50 Years Old) Lots 1-3 | Fluzone® (≥50 Years Old) | Total VCIV - Modified Manufacturing Process (All Participants) Lots 1-3 | Fluzone® (All Participants)
Number analyzed (Participants) | 598 | 201 | 201 | 594 | 203 | 1192 | 404
percentage of participants | 37.0 [33.1 to 41.0] | 44.3 [37.3 to 51.4] | 39.8 [33.0 to 46.9] | 19.5 [16.4 to 22.9] | 27.1 [21.1 to 33.8] | 28.3 [25.7 to 30.9] | 33.4 [28.8 to 38.2]

6. Secondary Outcome: Percentage of Participants With Injection Site Reactions
Time Frame: within 7 days post vaccination
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total VCIV - Modified Manufacturing Process (18-49 Year Old) Lots 1-3; Total VCIV - Modified Manufacturing Process (≥50 Year Old) Lots 1-3; Total VCIV - Modified Manufacturing Process (All Participants) Lots 1-3: Vero cell-derived trivalent influenza vaccine (VCIV)
  Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- VCIV Manufactured With Current Process (18-49 Year Old): Vero cell-derived trivalent influenza vaccine (VCIV)
  VCIV manufactured with the current manufacturing process (VCIV current)
- Fluzone® (18-49 Year Old): Fluzone®, licensed trivalent influenza vaccine (TIV)
  Fluzone®, licensed trivalent influenza vaccine (TIV)
Arm/Group | Total VCIV - Modified Manufacturing Process (18-49 Year Old) Lots 1-3 | VCIV Manufactured With Current Process (18-49 Year Old) | Fluzone® (18-49 Year Old) | Total VCIV - Modified Manufacturing Process (≥50 Year Old) Lots 1-3 | Fluzone® (≥50 Years Old) | Total VCIV - Modified Manufacturing Process (All Participants) Lots 1-3 | Fluzone® (All Participants)
Number analyzed (Participants) | 598 | 201 | 201 | 594 | 203 | 1192 | 404
percentage of participants | 50.7 [46.6 to 54.7] | 51.7 [44.6 to 58.8] | 44.3 [37.3 to 51.4] | 28.6 [25.0 to 32.4] | 30.5 [24.3 to 37.4] | 39.7 [36.9 to 42.5] | 37.4 [32.6 to 42.3]

7. Secondary Outcome: Number and Severity of Each Solicited Systemic Reaction and Injection Site Reaction
Time Frame: within 7 days post vaccination
Population: as for outcome 5
Measure: Number; unit: number of adverse reactions
Groups:
- VCIV - Modified Manufacturing Process (All Ages) Lots 1-3: Vero cell-derived trivalent influenza vaccine (VCIV)
  Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
- VCIV Manufactured With Current Process (All Ages): Vero cell-derived trivalent influenza vaccine (VCIV)
  VCIV manufactured with the current manufacturing process (VCIV current)
- Fluzone® (All Ages): Fluzone®, licensed trivalent influenza vaccine (TIV)
Arm/Group | Total VCIV - Modified Process (18 - 49 Years Old) Lots 1-3 | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | Total VCIV - Modified Process (≥50 Years Old) Lots 1-3 | Fluzone® (≥50 Years Old) | VCIV - Modified Manufacturing Process (All Ages) Lots 1-3 | VCIV Manufactured With Current Process (All Ages) | Fluzone® (All Ages)
Number analyzed (Participants) | 598 | 201 | 201 | 594 | 203 | 1192 | 201 | 404
number of adverse reactions
  Injection site redness- Mild | 5 | 2 | 1 | 11 | 3 | 16 | 2 | 4
  Injection site redness-Moderate | 2 | 0 | 1 | 2 | 0 | 4 | 0 | 1
  Injection site redness-Unknown | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1
  Injection site redness-Severe | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Injection site redness-Total | 9 | 2 | 2 | 14 | 4 | 23 | 2 | 6
  Injection site swelling-Mild | 5 | 0 | 1 | 7 | 1 | 12 | 0 | 2
  Injection site swelling-Moderate | 2 | 1 | 0 | 3 | 2 | 5 | 1 | 2
  Injection site sweling-Unknown | 1 | 0 | 0 | 2 | 1 | 3 | 0 | 1
  Injection site swelling-Total | 8 | 1 | 1 | 12 | 4 | 20 | 1 | 5
  Injection site induration-Mild | 5 | 3 | 1 | 8 | 1 | 13 | 3 | 1
  Injection site induration-Moderate | 6 | 1 | 1 | 3 | 1 | 9 | 1 | 2
  Injection site induration-Unknown | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 2
  Injection site induration-Total | 11 | 4 | 3 | 13 | 2 | 24 | 4 | 5
  Injection site pain-Mild | 174 | 67 | 50 | 67 | 20 | 241 | 67 | 70
  Injection site pain-Moderate | 6 | 1 | 0 | 6 | 1 | 12 | 1 | 1
  Injection site pain-Total | 180 | 68 | 50 | 73 | 21 | 253 | 68 | 71
  Injection site tenderness-Mild | 230 | 81 | 68 | 129 | 47 | 359 | 81 | 115
  Injection site tenderness-Moderate | 4 | 0 | 2 | 5 | 2 | 9 | 0 | 4
  Injection site tenderness-Total | 234 | 81 | 70 | 134 | 49 | 368 | 81 | 119
  Injection site ecchymosis-Mild | 23 | 6 | 4 | 8 | 5 | 31 | 6 | 9
  Injection site ecchymosis-Moderate | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
  Injection site ecchymosis-Total | 23 | 6 | 4 | 9 | 6 | 32 | 6 | 10
  Malaise-Mild | 86 | 42 | 32 | 49 | 16 | 135 | 42 | 48
  Malaise-Moderate | 22 | 10 | 8 | 10 | 3 | 32 | 10 | 11
  Malaise-Severe | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Malaise-Total | 108 | 52 | 40 | 60 | 19 | 168 | 52 | 59
  Shivering-Mild | 14 | 7 | 5 | 3 | 4 | 17 | 7 | 9
  Shivering-Moderate | 6 | 5 | 4 | 2 | 1 | 8 | 5 | 5
  Shivering-Severe | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Shivering-Total | 20 | 12 | 9 | 6 | 5 | 26 | 12 | 14
  Fatigue-Mild | 77 | 33 | 25 | 37 | 20 | 114 | 33 | 45
  Fatigue-Moderate | 28 | 9 | 10 | 18 | 5 | 46 | 9 | 15
  Fatigue-Severe | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1
  Fatigue-Total | 105 | 43 | 36 | 56 | 25 | 161 | 43 | 61
  Headache-Mild | 92 | 32 | 24 | 41 | 19 | 133 | 32 | 43
  Headache-Moderate | 17 | 7 | 9 | 8 | 6 | 25 | 7 | 15
  Headache-Severe | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Headache-Total | 109 | 39 | 33 | 50 | 25 | 159 | 39 | 58
  Sweating-Mild | 15 | 8 | 4 | 14 | 7 | 29 | 8 | 11
  Sweating-Moderate | 8 | 3 | 3 | 3 | 1 | 11 | 3 | 4
  Sweating-Severe | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Sweating-Total | 23 | 11 | 7 | 18 | 8 | 41 | 11 | 15
  Muscle pain-Mild | 85 | 34 | 26 | 53 | 17 | 138 | 34 | 43
  Muscle pain-Moderate | 16 | 6 | 12 | 8 | 3 | 24 | 6 | 15
  Muscle pain-Severe | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0
  Muscle pain-Total | 101 | 42 | 38 | 62 | 20 | 163 | 42 | 58
  Arthralgia (joint pain)-Mild | 30 | 5 | 4 | 10 | 6 | 40 | 5 | 10
  Arthralgia (joint pain)-Moderate | 6 | 4 | 3 | 6 | 1 | 12 | 4 | 4
  Arthralgia (joint pain)-Severe | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
  Arthralgia (joint pain)-Total | 36 | 9 | 8 | 17 | 7 | 53 | 9 | 15
  Nausea-Mild | 24 | 10 | 8 | 14 | 4 | 38 | 10 | 12
  Nausea-Moderate | 11 | 4 | 3 | 2 | 1 | 13 | 4 | 4
  Nausea-Severe | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Nausea-Total | 36 | 14 | 11 | 16 | 5 | 52 | 14 | 16
  Vomiting-Mild | 2 | 0 | 2 | 1 | 1 | 3 | 0 | 3
  Vomiting-Moderate | 6 | 1 | 2 | 0 | 0 | 6 | 1 | 2
  Vomiting-Severe | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Vomiting-Total | 9 | 1 | 4 | 1 | 1 | 10 | 1 | 5

8. Primary Outcome: Non-inferiority of Modified Manufacturing Process Compared to the Current Process
Description: Non-inferiority of modified manufacturing process compared to the current process.
  Co-primary analysis of HIA Titer for each of the three antigens (Outcome Measure 1) was performed on a subset of the Per Protocol analysis dataset for participants 18-49 Years Old treated with Vero cell-derived trivalent influenza vaccine (VCIV) from the modified manufacturing process and VCIV manufactured with the current process
Time Frame: 21 days post vaccination
Population: Subset of the per-protocol (PP) analysis dataset of Cohort 1 (18-49 years) comprising subjects from the VCIV modified and VCIV current treatment groups (because the aim of the analysis was to show non-inferiority between the two VCIV manufacturing processes), for all three strains separately.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio of Geometric Mean- no units
Groups:
- Strain A/H1N1: Strain A/H1N1 from the Vero cell-derived trivalent influenza vaccine (VCIV)
- Strain A/H3N2: Strain A/H3N2 from the Vero cell-derived trivalent influenza vaccine (VCIV)
- Strain B: Strain B from the Vero cell-derived trivalent influenza vaccine (VCIV)
Arm/Group | Strain A/H1N1 | Strain A/H3N2 | Strain B
Number analyzed (Participants) | 774 | 774 | 774
ratio of Geometric Mean- no units | 1.12 [0.93 to 1.35] | 1.16 [0.97 to 1.38] | 1.33 [1.11 to 1.60]
Statistical Analysis 1: Comparison: Strain A/H1N1 vs Strain A/H3N2 vs Strain B; Test type: Non-Inferiority or Equivalence — The probability that the modified process is noninferior to the current one (i.e. lower limit of the 95% CI of the ratio of geometric means [modified vs. current] is greater than or equal to 0.67) is above 99% for one strain, and it is around 97% for all three strains (considering the three strains to be independent, 0.99 x 0.99 x 0.99=0.97); ANCOVA = 0.67, 95% CI 1-sided [lower limit 0.67]

9. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: within 21 days post vaccination
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Total VCIV - Modified Process (18 - 49 Years Old) Lots 1-3 | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | Total VCIV - Modified Process (≥50 Years Old) Lots 1-3 | Fluzone® (≥50 Years Old)
Number analyzed (Participants) | 598 | 201 | 201 | 594 | 203
percentage of participants
  Serious AEs | 0.2 | 0 | 0 | 0.7 | 0
  Any non-serious systemic AEs | 47.7 | 53.2 | 48.3 | 35.4 | 38.4
  Treatment-related non-serious systemic AEs | 38.5 | 44.8 | 40.3 | 21.4 | 27.6
  Any non-serious local AEs | 50.8 | 51.7 | 44.3 | 28.8 | 31.5

10. Primary Outcome: Lot Consistency of the Three Modified Manufacturing Process Lots
Description: Lot consistency of the three modified manufacturing process lots Co-primary analysis of HIA Titer for each of the three antigens (Outcome Measure 1) was performed on a subset of the Per Protocol Analysis Dataset for participants of all ages treated with three Vero cell-derived trivalent influenza vaccine (VCIV) lots manufactured from the modified process.
Time Frame: 21 days post vaccination
Population: Subset of the PP analysis dataset comprising the 3 VCIV modified lots (as the aim of the analysis was to show similarity between three different lots of the VCIV manufactured with the modified process), both cohort pooled, for all three strains separately.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio of geometric mean- no units
Arm/Group | Strain A/H1N1 | Strain A/H3N2 | Strain B
Number analyzed (Participants) | 1163 | 1163 | 1163
ratio of geometric mean- no units
  Lot 2 vs. Lot 1 | 1.00 [0.84 to 1.19] | 1.15 [0.98 to 1.35] | 0.87 [0.74 to 1.03]
  Lot 3 vs. Lot 1 | 0.90 [0.76 to 1.07] | 1.17 [1.00 to 1.38] | 0.84 [0.71 to 0.99]
  Lot 3 vs. Lot 2 | 0.89 [0.75 to 1.06] | 1.02 [0.87 to 1.20] | 0.96 [0.81 to 1.13]
Statistical Analysis 1: Comparison: Strain A/H1N1 vs Strain A/H3N2 vs Strain B; The overall power to prove the similarity between the three lots for all three strains is approximately 99%. For the two primary co-analyses (Noninferiority and Lot Consistency), the overall power of the immunogenicity analyses is approximately 96% (calculated as 0.97 x 0.99=0.96); Test type: Superiority or Other; ANCOVA = 0.67, 95% CI 2-sided [0.67 to 1.5]

11. Primary Outcome: Percentage of Participants With Fever
Description: Percentage of participants with fever
Time Frame: onset within 7 days post vaccination
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants with fever
Groups:
- VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1-3: Vero cell-derived trivalent influenza vaccine (VCIV)
  Vero cell-derived trivalent influenza vaccine manufactured with the modified manufacturing process (VCIV modified)
Arm/Group | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 1 | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 2 | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 3 | Total VCIV - Modified Manufacturing Process (18-49 Years Old) Lots 1-3 | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1 | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 2 | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 3 | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1-3 | Fluzone® (≥50 Years Old)
Number analyzed (Participants) | 200 | 199 | 199 | 598 | 201 | 201 | 199 | 197 | 198 | 594 | 203
percentage of participants with fever | 2.5 [0.8 to 5.7] | 1.0 [0.1 to 3.6] | 2.0 [0.6 to 5.1] | 1.8 [0.9 to 3.3] | 1.0 [0.1 to 3.5] | 0.0 [0.0 to 1.8] | 2.5 [0.8 to 5.8] | 1.0 [0.1 to 3.6] | 2.0 [0.6 to 5.1] | 1.9 [0.9 to 3.3] | 0.0 [0.0 to 1.8]
Statistical Analysis 1: Comparison: Total VCIV - Modified Manufacturing Process (18-49 Years Old) Lots 1-3 vs Fluzone® (18-49 Years Old); Test type: Non-Inferiority or Equivalence — Differences between fever incidences (95% CI) between treatment groups VCIV Modified (Total) and TIV was computed for each age cohort separately. The Confidence Interval estimation method was the method of Miettinen & Nurminen, as described in the StatXact User Manual (i.e. the score statistics, also called Chan's method, page 283). Noninferiority will be concluded if the upper limit of the 95% CI (VCIV modified-TIV) is <5%; Method of Miettinen & Nurminen = 1.8, 95% CI [0.1 to 3.3]

12. Secondary Outcome: Frequency and Severity of Related Adverse Events
Description: Frequency and severity of adverse events considered related to the vaccination (possibly related, probably related, unknown) according to System Organ Class (SOC) and Preferred Term (PT) SOCs are abbreviated as follows:- BLD- Blood and lymphatic system disorders EAR- Ear and labyrinth disorders EYE- Eye disorders GID- Gastrointestinal disorders GEN- General disorders and administration site conditions IMM- Immune system disorders INF- Infections and infestations MET- Metabolism and nutrition disorders MSK- Musculoskeletal and connective tissue disorders NER- Nervous system disorders RES- Respiratory, thoracic and mediastinal disorders SKN- Skin and subcutaneous tissue disorders VAS- Vascular disorders
  SYS-Systemic LOC-Local
Time Frame: within 21 days post vaccination
Population: as for outcome 5
Measure: Number; unit: percentage of related adverse events
Arm/Group | Total VCIV - Modified Process (18 - 49 Years Old) Lots 1-3 | VCIV Manufactured With Current Process (18-49 Years Old) | Fluzone® (18-49 Years Old) | Total VCIV - Modified Process (≥50 Years Old) Lots 1-3 | Fluzone® (≥50 Years Old)
Number analyzed (Participants) | 598 | 201 | 201 | 594 | 203
percentage of related adverse events
  LOC-GEN-Injection Site Anaesthesia-Mild | 0 | 0 | 0.5 | 0 | 0
  LOC-GEN-Injection Site Anaesthesia-Total | 0 | 0 | 0.5 | 0 | 0
  LOC-GEN-Injection Site Bruising-Mild | 0 | 0.5 | 0 | 0 | 0
  LOC-GEN-Injection Site Bruising-Total | 0 | 0.5 | 0 | 0 | 0
  LOC-GEN-Injection Site Discolouration-Mild | 0 | 0 | 0 | 0.5 | 0
  LOC-GEN-Injection Site Discolouration-Total | 0 | 0 | 0 | 0.5 | 0
  LOC-GEN-Injection Site Erythema-Mild | 0.8 | 1.0 | 0.5 | 1.9 | 1.5
  LOC-GEN-Injection Site Erythema-Moderate | 0.3 | 0 | 0.5 | 0.3 | 0
  LOC-GEN-Injection Site Erythema-Severe | 0.2 | 0 | 0 | 0 | 0
  LOC-GEN-Injection Site Erythema-Unknown | 0.2 | 0 | 0 | 0.2 | 0.5
  LOC-GEN-Injection Site Erythema-Total | 1.5 | 0 | 0 | 0 | 0
  LOC-GEN-Injection Site Exfoliation-Mild | 0.2 | 0 | 0 | 0 | 0
  LOC-GEN-Injection Site Exfoliation-Total | 0.2 | 0 | 0 | 0 | 0
  LOC-GEN-Injection Site Haemorrhage-Mild | 3.8 | 3.0 | 2.0 | 1.3 | 2.5
  LOC-GEN-Injection Site Haemorrhage-Moderate | 0 | 0 | 0 | 0.2 | 0.5
  LOC-GEN-Injection Site Haemorrhage-Total | 3.8 | 0 | 0 | 0 | 0
  LOC-GEN-Injection Site Induration-Mild | 0.8 | 1.5 | 0.5 | 1.3 | 0
  LOC-GEN-Injection Site Induration-Moderate | 1.0 | 0.5 | 0.5 | 0.5 | 0.5
  LOC-GEN-Injection Site Induration-Unknown | 0 | 0 | 0 | 0.3 | 0.5
  LOC-GEN-Injection Site Induration-Total | 0 | 0 | 0 | 2.2 | 1.0
  LOC-GEN-Injection Site Pain-Mild | 47.5 | 50.2 | 42.3 | 25.1 | 26.6
  LOC-GEN-Injection Site Pain-Moderate | 1.3 | 0.5 | 1.0 | 1.2 | 1.0
  LOC-GEN-Injection Site Pain-Total | 48.8 | 0 | 0 | 0 | 0
  LOC-GEN-Injection Site Pruritus-Mild | 1.0 | 0 | 0.5 | 0.7 | 0.5
  LOC-GEN-Injection Site Pruritus-Moderate | 0 | 0 | 0.5 | 0 | 0
  LOC-GEN-Injection Site Pruritus-Total | 1.0 | 0 | 0 | 0 | 0
  LOC-GEN-Injection Site Rash-Mild | 0 | 0.5 | 0 | 0.2 | 0
  LOC-GEN-Injection Site Rash-Total | 0 | 0.5 | 0 | 0.2 | 0
  LOC-GEN-Injection Site Reaction-Mild | 0.7 | 0 | 0 | 0.2 | 0.5
  LOC-GEN-Injection Site Reaction-Total | 0.7 | 0 | 0 | 0.2 | 0.5
  LOC-GEN-Injection Site Scab-Mild | 0.2 | 0 | 0 | 0 | 0.5
  LOC-GEN-Injection Site Scab-Total | 0.2 | 0 | 0 | 0 | 0.5
  LOC-GEN-Injection Site Swelling-Mild | 0.8 | 0 | 0.5 | 1.2 | 0.5
  LOC-GEN-Injection Site Swelling-Moderate | 0.3 | 0.5 | 0 | 0.5 | 1.0
  LOC-GEN-Injection Site Swelling-Unknown | 0.2 | 0 | 0 | 0.3 | 0.5
  LOC-GEN-Injection Site Swelling-Total | 1.3 | 0 | 0 | 2.0 | 2.0
  LOC-GEN-Injection Site Warmth-Mild | 0.2 | 1.0 | 0 | 0.2 | 0
  LOC-GEN-Injection Site Warmth-Total | 0.2 | 1.0 | 0 | 0.2 | 0
  LOC-GEN-MILD-TOTAL | 48.5 | 50.7 | 41.8 | 25.9 | 29.1
  LOC-GEN-MODERATE-TOTAL | 1.8 | 1.0 | 2.0 | 2.2 | 2.0
  LOC-GEN-SEVERE-TOTAL | 0.2 | 0 | 0 | 0 | 0
  LOC-GEN-UNKNOWN-TOTAL | 0.3 | 0 | 0.5 | 0.7 | 0.5
  LOC-GEN-TOTAL | 50.8 | 51.7 | 44.3 | 28.8 | 31.5
  SYS-BLD-Lymph node pain-Mild | 0 | 0 | 0 | 0.2 | 0
  SYS-BLD-Lymph node pain-Total | 0 | 0 | 0 | 0.2 | 0
  SYS-BLD-Lymphadenopathy-Mild | 0.3 | 0 | 0 | 0 | 0
  SYS-BLD-Lymphadenopathy-Moderate | 0.2 | 0 | 0 | 0 | 0
  SYS-BLD-Lymphadenopathy-Total | 0.5 | 0 | 0 | 0 | 0
  SYS-BLD-MILD-TOTAL | 0.3 | 0 | 0 | 0.2 | 0
  SYS-BLD-MODERATE-TOTAL | 0.2 | 0 | 0 | 0 | 0
  SYS-BLD-TOTAL | 0.5 | 0 | 0 | 0.2 | 0
  SYS-EAR-Ear pain-Mild | 0.2 | 0.5 | 0 | 0 | 0
  SYS-EAR-Ear pain-Total | 0.2 | 0.5 | 0 | 0 | 0
  SYS-EAR-MILD-TOTAL | 0.2 | 0.5 | 0 | 0 | 0
  SYS-EAR-TOTAL | 0.2 | 0.5 | 0 | 0 | 0
  SYS-EYE-Dark circles under eyes-Mild | 0 | 0 | 0 | 0.2 | 0
  SYS-EYE-Dark circles under eyes-Total | 0 | 0 | 0 | 0.2 | 0
  SYS-EYE-Eye pruritus-Mild | 0 | 0.5 | 0 | 0.2 | 0
  SYS-EYE-Eye pruritus-Total | 0 | 0.5 | 0 | 0.2 | 0
  SYS-EYE-MILD-TOTAL | 0 | 0.5 | 0 | 0.3 | 0
  SYS-EYE-TOTAL | 0 | 0.5 | 0 | 0.3 | 0
  SYS-GID-Abdominal pain upper-Moderate | 0 | 0 | 0 | 0 | 0.5
  SYS-GID-Abdominal pain upper-Total | 0 | 0 | 0 | 0 | 0.5
  SYS-GID-Apthous stomatitis-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-GID-Apthous stomatitis-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-GID-Diarrhoea-Mild | 0.5 | 0 | 0 | 0.2 | 0
  SYS-GID-Diarrhoea-Moderate | 0.3 | 0 | 0 | 0 | 0
  SYS-GID-Diarrhoea-Total | 0.8 | 0 | 0 | 0.2 | 0
  SYS-GID-Hypoaesthesia oral-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-GID-Hypoaesthesia oral-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-GID-Nausea-Mild | 3.8 | 5.0 | 3.0 | 2.2 | 2.0
  SYS-GID-Nausea-Moderate | 1.8 | 2.0 | 1.5 | 0.3 | 0.5
  SYS-GID-Nausea-Severe | 0.2 | 0 | 0 | 0 | 0
  SYS-GID-Nausea-Total | 5.9 | 7.0 | 4.5 | 2.5 | 2.5
  SYS-GID-Oedema mouth-Mild | 0 | 0.5 | 0 | 0 | 0
  SYS-GID-Oedema mouth-Total | 0 | 0.5 | 0 | 0 | 0
  SYS-GID-Vomiting-Mild | 0.3 | 0 | 1.0 | 0.2 | 0.5
  SYS-GID-Vomiting-Moderate | 1.0 | 0.5 | 1.0 | 0 | 0
  SYS-GID-Vomiting-Severe | 0.2 | 0 | 0 | 0 | 0
  SYS-GID-Vomiting-Total | 1.5 | 0.5 | 2.0 | 0.2 | 0.5
  SYS-GID-MILD-TOTAL | 4.0 | 5.0 | 3.0 | 2.4 | 2.0
  SYS-GID-MODERATE-TOTAL | 2.2 | 2.0 | 2.0 | 0.3 | 1.0
  SYS-GID-SEVERE-TOTAL | 0.2 | 0 | 0 | 0 | 0
  SYS-GID-TOTAL | 6.4 | 7.0 | 5.0 | 2.7 | 3.0
  SYS-GEN-Chest discomfort-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Chest discomfort-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Chest pain-Mild | 0 | 0.5 | 0 | 0 | 0
  SYS-GEN-Chest pain-Total | 0 | 0.5 | 0 | 0 | 0
  SYS-GEN-Chills-Mild | 2.5 | 3.5 | 2.0 | 0.5 | 2.5
  SYS-GEN-Chills-Moderate | 1.0 | 2.5 | 2.0 | 0.3 | 0.5
  SYS-GEN-Chills-Severe | 0 | 0 | 0 | 0.2 | 0
  SYS-GEN-Chills-Total | 3.5 | 6.0 | 4.0 | 1.0 | 3.0
  SYS-GEN-Discomfort-Mild | 0.2 | 1.0 | 0 | 0.2 | 0
  SYS-GEN-Discomfort-Total | 0.2 | 1.0 | 0 | 0.2 | 0
  SYS-GEN-Fatigue-Mild | 12 | 14.9 | 10.9 | 5.6 | 9.4
  SYS-GEN-Fatigue-Moderate | 4.5 | 4.5 | 5.0 | 2.9 | 2.5
  SYS-GEN-Fatigue-Severe | 0 | 0.5 | 0.5 | 0.2 | 0
  SYS-GEN-Fatigue-Total | 16.6 | 19.9 | 16.4 | 8.6 | 11.8
  SYS-GEN-Feeling abnormal-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Feeling abnormal-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Feeling cold-Mild | 0 | 0 | 0 | 0.2 | 0.5
  SYS-GEN-Feeling cold-Total | 0 | 0 | 0 | 0.2 | 0.5
  SYS-GEN-Injection site pain-Mild | 0.2 | 0 | 0 | 0.2 | 0
  SYS-GEN-Injection site pain-Total | 0.2 | 0 | 0 | 0.2 | 0
  SYS-GEN-Injection site reaction-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Injection site reaction-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Malaise-Mild | 14.4 | 20.9 | 15.9 | 7.7 | 7.4
  SYS-GEN-Malaise-Moderate | 3.5 | 5.0 | 4.0 | 1.7 | 1.5
  SYS-GEN-Malaise-Severe | 0 | 0 | 0 | 0.2 | 0
  SYS-GEN-Malaise-Total | 17.9 | 25.9 | 19.9 | 9.6 | 8.9
  SYS-GEN-Nodule-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Nodule-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Non-cardiac chest pain-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Non-cardiac chest pain-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-GEN-Oedema peripheral-Moderate | 0 | 0 | 0 | 0 | 0.5
  SYS-GEN-Oedema peripheral-Total | 0 | 0 | 0 | 0 | 0.5
  SYS-GEN-Pain-Mild | 0.3 | 1.0 | 0.5 | 0.3 | 0
  SYS-GEN-Pain-Moderate | 0.2 | 0 | 0 | 0.3 | 0
  SYS-GEN-Pain-Total | 0.5 | 1.0 | 0.5 | 0.7 | 0
  SYS-GEN-Pyrexia-Mild | 1.3 | 0.5 | 0 | 1.0 | 0.5
  SYS-GEN-Pyrexia-Moderate | 0.3 | 0 | 0 | 0.2 | 0
  SYS-GEN-Pyrexia-Severe | 0.2 | 0.5 | 0 | 0.2 | 0
  SYS-GEN-Pyrexia-Total | 1.8 | 1.0 | 0 | 1.3 | 0.5
  SYS-GEN-MILD-TOTAL | 20.6 | 26.4 | 22.9 | 10.4 | 13.8
  SYS-GEN-MODERATE-TOTAL | 6.7 | 8.5 | 6.5 | 3.5 | 3.9
  SYS-GEN-SEVERE-TOTAL | 0.2 | 1.0 | 0.5 | 0.3 | 0
  SYS-GEN-TOTAL | 27.4 | 35.8 | 29.9 | 14.3 | 17.7
  SYS-INF-Acute sinusitis-Moderate | 0.2 | 0 | 0 | 0 | 0
  SYS-INF-Acute sinusitis-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-INF-Herpes simplex-Moderate | 0.2 | 0 | 0 | 0 | 0
  SYS-INF-Herpes simplex-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-INF-Nasopharyngitis-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-INF-Nasopharyngitis-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-INF-Oral herpes-Mild | 0 | 0.5 | 0 | 0 | 0
  SYS-INF-Oral herpes-Total | 0 | 0.5 | 0 | 0 | 0
  SYS-INF-Otitis media-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-INF-Otitis media-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-INF-Sinusitis-Mild | 0.3 | 0 | 0 | 0 | 0
  SYS-INF-Sinusitis-Total | 0.3 | 0 | 0 | 0 | 0
  SYS-INF-Upper respiratory tract infection-Mild | 0 | 0 | 0 | 0.2 | 0
  SYS-INF-Upper respiratory tract infection-Moderate | 0 | 0 | 0 | 0.2 | 0
  SYS-INF-Upper respiratory tract infection-Total | 0 | 0 | 0 | 0.3 | 0
  SYS-INF-MILD-TOTAL | 0.7 | 0.5 | 0 | 0.2 | 0
  SYS-INF-MODERATE-TOTAL | 0.3 | 0 | 0 | 0.2 | 0
  SYS-INF-TOTAL | 1.0 | 0.5 | 0 | 0.3 | 0
  SYS-MET-Decreased appetite-Mild | 0 | 0 | 0 | 0.2 | 0
  SYS-MET-Decreased appetite-Total | 0 | 0 | 0 | 0.2 | 0
  SYS-MET-MILD-TOTAL | 0 | 0 | 0 | 0.2 | 0
  SYS-MET-TOTAL | 0 | 0 | 0 | 0.2 | 0
  SYS-MSK-Arthralgia-Mild | 4.5 | 2.5 | 2.0 | 1.5 | 3.0
  SYS-MSK-Arthralgia-Moderate | 1.0 | 2.0 | 1.5 | 1.0 | 0.5
  SYS-MSK-Arthralgia-Severe | 0 | 0 | 0.5 | 0.2 | 0
  SYS-MSK-Arthralgia-Total | 5.5 | 4.5 | 4.0 | 2.7 | 3.4
  SYS-MSK-Back pain-Mild | 0.2 | 0.5 | 0 | 0.5 | 0
  SYS-MSK-Back pain-Moderate | 0 | 0 | 0.5 | 0 | 0
  SYS-MSK-Back pain-Total | 0.2 | 0.5 | 0.5 | 0.5 | 0
  SYS-MSK-Joint swelling-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-MSK-Joint swelling-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-MSK-Muscle spasms-Mild | 0 | 0.5 | 0 | 0.2 | 0
  SYS-MSK-Muscle spasms-Moderate | 0 | 0 | 0 | 0.2 | 0
  SYS-MSK-Muscle spasms-Total | 0 | 0.5 | 0 | 0.3 | 0
  SYS-MSK-Muscle tightness-Mild | 0.3 | 0 | 0 | 0 | 0
  SYS-MSK-Muscle tightness-Total | 0.3 | 0 | 0 | 0 | 0
  SYS-MSK-Musculoskeletal pain-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-MSK-Musculoskeletal pain-Moderate | 0 | 0 | 0 | 0.2 | 0
  SYS-MSK-Musculoskeletal pain-Total | 0.2 | 0 | 0 | 0.2 | 0
  SYS-MSK-Musculoskeletal stiffness-Mild | 0.3 | 0 | 0 | 0 | 0.5
  SYS-MSK-Musculoskeletal stiffness-Total | 0.3 | 0 | 0 | 0 | 0.5
  SYS-MSK-Myalgia-Mild | 13.7 | 15.9 | 11.9 | 8.6 | 8.4
  SYS-MSK-Myalgia-Moderate | 2.5 | 3.0 | 6.0 | 1.3 | 1.5
  SYS-MSK-Myalgia-Severe | 0 | 1.0 | 0 | 0.2 | 0
  SYS-MSK-Myalgia-Total | 16.2 | 19.9 | 17.9 | 10.1 | 9.9
  SYS-MSK-Neck pain-Mild | 0.3 | 0 | 0 | 0 | 0
  SYS-MSK-Neck pain-Total | 0.3 | 0 | 0 | 0 | 0
  SYS-MSK-Pain in extremity-Mild | 0 | 0 | 0.5 | 0.3 | 0.5
  SYS-MSK-Pain in extremity-Total | 0 | 0 | 0.5 | 0.3 | 0.5
  SYS-MSK-Pain in jaw-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-MSK-Pain in jaw-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-MSK-MILD-TOTAL | 14.7 | 16.9 | 12.4 | 9.3 | 10.8
  SYS-MSK-MODERATE-TOTAL | 2.7 | 3.5 | 5.5 | 1.3 | 1.5
  SYS-MSK-SEVERE-TOTAL | 0 | 1.0 | 0.5 | 0.2 | 0
  SYS-MSK-TOTAL | 17.4 | 21.4 | 18.4 | 10.8 | 12.3
  SYS-NER-Burning sensation-Mild | 0 | 0 | 0 | 0.2 | 0
  SYS-NER-Burning sensation-Total | 0 | 0 | 0 | 0.2 | 0
  SYS-NER-Dizziness-Mild | 0.3 | 0.5 | 0 | 0.2 | 0
  SYS-NER-Dizziness-Total | 0.3 | 0.5 | 0 | 0.2 | 0
  SYS-NER-Dysgeusia-Mild | 0 | 0.5 | 0 | 0 | 0
  SYS-NER-Dysgeusia-Moderate | 0 | 0 | 0 | 0 | 0.5
  SYS-NER-Dysgeusia-Total | 0 | 0.5 | 0 | 0 | 0.5
  SYS-NER-Headache-Mild | 13.4 | 13.4 | 10.9 | 6.1 | 7.9
  SYS-NER-Headache-Moderate | 3.0 | 3.5 | 4.5 | 1.2 | 3.0
  SSYS-NER-Headache-Severe | 0 | 0 | 0 | 0.2 | 0
  SYS-NER-Headache-Total | 16.4 | 16.9 | 15.4 | 7.4 | 10.8
  SYS-NER-Hypoaesthesia-Mild | 0.3 | 0 | 0 | 0 | 0
  SYS-NER-Hypoaesthesia-Total | 0.3 | 0 | 0 | 0 | 0
  SYS-NER-Lethargy-Mild | 0 | 0.5 | 0 | 0 | 0
  SYS-NER-Lethargy-Total | 0 | 0.5 | 0 | 0 | 0
  SYS-NER-Paraesthesia-Mild | 0.3 | 0 | 0 | 0 | 0
  SYS-NER-Paraesthesia-Total | 0.3 | 0 | 0 | 0 | 0
  SYS-NER-Sinus headache-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-NER-Sinus headache-Moderate | 0.2 | 0 | 0 | 0 | 0
  SYS-NER-Sinus headache-Total | 0.3 | 0 | 0 | 0 | 0
  SYS-NER-MILD-TOTAL | 13.4 | 13.9 | 10.9 | 6.4 | 7.9
  SYS-NER-MODERATE-TOTAL | 3.2 | 3.5 | 4.5 | 1.2 | 3.0
  SYS-NER-SEVERE-TOTAL | 0 | 0 | 0 | 0.2 | 0
  SYS-NER-TOTAL | 16.6 | 17.4 | 15.4 | 7.7 | 10.8
  SYS-RES-Cough-Mild | 0.7 | 0.5 | 0.5 | 0.2 | 0.5
  SYS-RES-Cough-Moderate | 0.7 | 0.5 | 0 | 0.2 | 0
  SYS-RES-Cough-Total | 1.3 | 1.0 | 0.5 | 0.3 | 0.5
  SYS-RES-Increased upper airway secretion-Mild | 0 | 0 | 0 | 0 | 0.5
  SYS-RES-Increased upper airway secretion-Moderate | 0 | 0 | 0 | 0.2 | 0
  SYS-RES-Increased upper airway secretion-Total | 0 | 0 | 0 | 0.2 | 0.5
  SYS-RES-Nasal congestion-Mild | 0.3 | 0.5 | 1.5 | 0.3 | 0
  SYS-RES-Nasal congestion-Moderate | 0.2 | 0 | 0 | 0.2 | 0.5
  SYS-RES-Nasal congestion-Total | 0.5 | 0.5 | 1.5 | 0.5 | 0.5
  SYS-RES-Oropharyngeal pain-Mild | 0.5 | 2.0 | 0 | 0.3 | 0.5
  SYS-RES-Oropharyngeal pain-Moderate | 0.8 | 0 | 0 | 0 | 0
  SYS-RES-Oropharyngeal pain-Total | 1.3 | 2.0 | 0 | 0.3 | 0.5
  SYS-RES-Paranasal sinus hypersecretion-Moderate | 0.2 | 0 | 0 | 0 | 0
  SYS-RES-Paranasal sinus hypersecretion-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-RES-Productive cough-Moderate | 0.2 | 0 | 0 | 0 | 0
  SYS-RES-Productive cough-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-RES-Respiratory tract congestion-Mild | 0.5 | 0 | 0 | 0.2 | 0
  SYS-RES-Respiratory tract congestion-Moderate | 0.2 | 0 | 0 | 0 | 0
  SYS-RES-Respiratory tract congestion-Total | 0.7 | 0 | 0 | 0.2 | 0
  SYS-RES-Rhinorrhoea-Mild | 1.0 | 0.5 | 0.5 | 0.3 | 0
  SYS-RES-Rhinorrhoea-Moderate | 0.3 | 0 | 0 | 0.2 | 0
  SYS-RES-Rhinorrhoea-Total | 1.3 | 0.5 | 0.5 | 0.5 | 0
  SYS-RES-Sinus congestion-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-RES-Sinus congestion-Moderate | 0.2 | 0 | 0 | 0 | 0
  SYS-RES-Sinus congestion-Total | 0.3 | 0 | 0 | 0 | 0
  SYS-RES-Sneezing-Mild | 0.7 | 0 | 0 | 0 | 0
  SYS-RES-Sneezing-Total | 0.7 | 0 | 0 | 0 | 0
  SYS-RES-Throat irritation-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-RES-Throat irritation-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-RES-MILD-TOTAL | 1.8 | 2.5 | 2.0 | 0.8 | 0.5
  SYS-RES-MODERATE-TOTAL | 1.5 | 0.5 | 0 | 0.3 | 0.5
  SYS-RES-TOTAL | 3.3 | 3.0 | 2.0 | 1.2 | 1.0
  SYS-SKN-Dermatitis allergic-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-SKN-Dermatitis allergic-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-SKN-Dermatitis contact-Mild | 0 | 0 | 0 | 0 | 0.5
  SYS-SKN-Dermatitis contact-Total | 0 | 0 | 0 | 0 | 0.5
  SYS-SKN-Erythema-Mild | 0 | 0.5 | 0 | 0 | 0
  SYS-SKN-Erythema-Total | 0 | 0.5 | 0 | 0 | 0
  SYS-SKN-Hyperhidrosis-Mild | 2.5 | 4.0 | 2.0 | 1.9 | 3.0
  SYS-SKN-Hyperhidrosis-Moderate | 1.3 | 1.5 | 1.5 | 0.5 | 0.5
  SYS-SKN-Hyperhidrosis-Severe | 0 | 0 | 0 | 0.2 | 0
  SYS-SKN-Hyperhidrosis-Total | 3.8 | 5.5 | 3.5 | 2.5 | 3.4
  SYS-SKN-Night sweats-Mild | 0 | 0 | 0 | 0.2 | 0
  SYS-SKN-Night sweats-Total | 0 | 0 | 0 | 0.2 | 0
  SYS-SKN-Pruritus-Mild | 0.2 | 0 | 0 | 0.2 | 0
  SYS-SKN-Pruritus-Total | 0.2 | 0 | 0 | 0.2 | 0
  SYS-SKN-Rash-Mild | 0.3 | 0 | 0 | 0.2 | 0
  SYS-SKN-Rash-Total | 0.3 | 0 | 0 | 0.2 | 0
  SYS-SKN-Skin mass-Mild | 0.2 | 0 | 0 | 0 | 0
  SYS-SKN-Skin mass-Total | 0.2 | 0 | 0 | 0 | 0
  SYS-SKN-MILD-TOTAL | 3.3 | 4.5 | 2.0 | 2.4 | 3.0
  SYS-SKN-MODERATE-TOTAL | 1.3 | 1.5 | 1.5 | 0.5 | 0.5
  SYS-SKN-SEVERE-TOTAL | 0 | 0 | 0 | 0.2 | 0
  SYS-SKN-TOTAL | 4.7 | 6.0 | 3.5 | 3.0 | 3.4
  SYS-VAS-Pallor-Mild | 0 | 0 | 0 | 0.2 | 0
  SYS-VAS-Pallor-Total | 0 | 0 | 0 | 0.2 | 0
  SYS-VAS-MILD-TOTAL | 0 | 0 | 0 | 0.2 | 0
  SYS-VAS-TOTAL | 0 | 0 | 0 | 0.2 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period of approximately 2.5 months
Groups:
- VCIV Manufactured With Current Process: Vero cell-derived trivalent influenza vaccine (VCIV)
  VCIV manufactured with the current manufacturing process (VCIV current)
- Fluzone® (18-49 Years Old); Fluzone® (≥50 Years Old): Fluzone®, licensed trivalent influenza vaccine (TIV) Fluzone®, licensed trivalent influenza vaccine (TIV)
Arm/Group | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 1 | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 2 | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 3 | VCIV Manufactured With Current Process | Fluzone® (18-49 Years Old) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1 | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 2 | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 3 | Fluzone® (≥50 Years Old)
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/199 | 0/199 | 0/201 | 0/201 | 0/199 | 0/197 | 0/198 | 0/203
Serious Adverse Events (participants affected / at risk) | 1/200 | 0/199 | 0/199 | 0/201 | 0/201 | 1/199 | 1/197 | 2/198 | 0/203
Other Adverse Events (participants affected / at risk) | 133/200 | 124/199 | 120/199 | 132/201 | 125/201 | 97/199 | 84/197 | 96/198 | 100/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 1 (N=200) | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 2 (N=199) | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 3 (N=199) | VCIV Manufactured With Current Process (N=201) | Fluzone® (18-49 Years Old) (N=201) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1 (N=199) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 2 (N=197) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 3 (N=198) | Fluzone® (≥50 Years Old) (N=203)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 1 (N=200) | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 2 (N=199) | VCIV - Modified Manufacturing Process (18-49 Years Old) Lot 3 (N=199) | VCIV Manufactured With Current Process (N=201) | Fluzone® (18-49 Years Old) (N=201) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 1 (N=199) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 2 (N=197) | VCIV - Modified Manufacturing Process (≥50 Years Old) Lot 3 (N=198) | Fluzone® (≥50 Years Old) (N=203)
Nausea (Gastrointestinal disorders) | 23 | 14 | 12 | 17 | 13 | 5 | 8 | 10 | 7
Chills (General disorders) | 13 | 4 | 7 | 14 | 11 | 4 | 7 | 4 | 6
Fatigue (General disorders) | 33 | 38 | 38 | 44 | 37 | 24 | 18 | 22 | 28
Malaise (General disorders) | 40 | 42 | 38 | 55 | 44 | 26 | 19 | 24 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 11 | 11 | 13 | 9 | 9 | 7 | 6 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 37 | 29 | 36 | 41 | 39 | 22 | 25 | 22 | 23
Headache (Nervous system disorders) | 50 | 43 | 39 | 44 | 41 | 25 | 21 | 18 | 27
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 4 | 12 | 4 | 3 | 2 | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 | 8 | 11 | 12 | 10 | 6 | 8 | 5 | 7
Injection site pain (General disorders) | 102 | 100 | 90 | 102 | 87 | 59 | 39 | 58 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements may vary with individual PIs, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or up to 18 months after study completion. Baxter requires a review of results communications (eg for confidential information) ≥60 days prior to submission/communication. Baxter may request additional delay of ≤60 days(e.g. for intellectual property protection). Prior authorization may be required.